CLINICAL TRIAL: NCT06258915
Title: Randomized Controlled Multicenter Study Comparing Efficacy and Safety of Adalimumab to That of Mycophenolate Mofetil in Steroid Dependent Non-infectious Uveitis
Brief Title: Treatment FOr Corticosteroid Dependent UveitiS
Acronym: FOCUS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP211032
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Non Infectious Uveitis
Keywords: Non-infectious uveitis; Macular oedema; Retinal vascularitis; Adalimumab; Mycophenolate mofetil
MeSH Terms: conditions — Macular Edema | interventions — Adalimumab; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab
- Mycophenolate mofetil (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Adalimumab — Adalimumab (80mg at day 0, then 40mg/14 days from W1 to W35 subcutaneously)
  Arms: Adalimumab
Drug: Mycophenolate Mofetil — 2 g/day orally for 36 weeks
  Arms: Mycophenolate mofetil

SUMMARY:
FOCUS is the first prospective randomized study comparing standard of care (mycophenolate mofetil) to adalimumab in recently active non infectious uveitis (NIU) with steroid dependency. There is no firm evidence or randomized trials that compared classical immunosuppressive compounds to biological agents; or identified the best treatment in this condition. The burden of NIU has been reduced with the use of immunosuppressive agents and biologics, raising the question of which of these compounds should be preferentially used in recently active NIU with steroid dependency.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to the performance of any study-specific procedures
2. ≥18 years of age
3. Diagnosis of non-infectious intermediate, posterior-, or pan-uveitis in at least one eye fulfilling the International Study Group Classification Criteria (Standardization of Uveitis Nomenclature [SUN] criteria) of posterior, or pan- uveitis confirmed by documented medical history
4. Recent activity of Non Infectious Uveitis as defined by the presence of at least 1 of the following parameters in either eye within the 3 months prior to inclusion visit despite >7mg/day of oral prednisone:

   * Active chorioretinal or retinal vascular lesion
   * Presence of macular edema by optical coherence.
   * ≥ 2+ anterior chamber cells (Standardization of Uveitis Nomenclature [SUN] criteria)
   * ≥ 2+ vitreous haze (National Eye Institute [NEI]/SUN criteria)
5. Chest X-ray (postero-anterior and lateral) or CT-scanner results within 12 weeks prior to inclusion with no evidence of active Tuberculosis, active infection, or malignancy
6. A potential subject with a positive interferon-gamma release assay (IGRA) (e.g., QuantiFERON®-TB Gold or T-spot TB® Test) at inclusion is eligible if:

   1. Her/his chest X-ray does not show evidence suggestive of active tuberculosis disease
   2. And there are no clinical signs and symptoms of pulmonary and/or extra-pulmonary tuberculosis disease.
   3. And these subjects with a latent tuberculosis infection who have not already received a prophylactic tuberculosis treatment must agree in advance to complete such a treatment course.
7. For female subjects of child-bearing potential: a negative pregnancy test at inclusion
8. For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study and 3 months and 5 months after stopping therapy for Mycophenolate mofetil (MMF) and adalimumab, respectively, unless sterility is confirmed. The simultaneous use of two complementary methods of contraception is preferable. Methods which may be considered as highly effective methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods (according to Clinical Trial Falicitation Group (CTFG) recommendations). Such methods include:

   For Female subjects :
   1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation 1:

      * oral
      * intravaginal
      * transdermal
   2. progestogen-only hormonal contraception associated with inhibition of ovulation:

      * oral
      * injectable
      * implantable
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system (IUS)
   5. bilateral tubal occlusion
   6. vasectomised partner
   7. sexual abstinence (In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject).

   For male subjects :
   1. use of condoms
   2. vasectomy (with documentation of azoospermia)
   3. sexual abstinence
9. Affiliated to a social security system

Exclusion Criteria:

1. Infectious uveitis, masquerade syndromes (idiopathic uveitis is permitted)
2. Isolated anterior uveitis
3. Monocular patient
4. Active tuberculosis
5. Positive HIV serology or Hepatitis C Virus (HCV) Hepatitis B Virus (HBV) Ag test
6. History of malignancy within 5 years prior to Inclusion other than carcinoma in situ of the cervix, non-metastatic squamous or basal cell carcinoma of the skin.
7. History of severe allergic or anaphylactic reactions to monoclonal antibodies, mycophenolate mofetil, rifampicin, isoniazid or fluorescein
8. Infection requiring treatment with intravenous antibiotics within 3 weeks prior to inclusion
9. History of multiple sclerosis and/or demyelinating disorder
10. Laboratory values assessed during inclusion:

    * Hemoglobin < 8g/dL
    * Whole Blood Count (WBC) < 2.0 x 103/mm3
    * Platelet count < 80 x 103/mm3
    * Glomerular filtration rates (GFR) <30ml/min.
    * Transaminases > 3 times upper normal value
11. Use of the following systemic treatments during the specified periods:

    * Treatment with any systemic alkylating agents within 12 months prior to inclusion (e.g., cyclophosphamide, chlorambucil)
    * Any live (attenuated) vaccine within 4 weeks prior to inclusion.
12. Stage III and IV New York Heart Association (NYHA) cardiac insufficiency
13. Pregnancy or breastfeeding
14. Under legal protection
15. Participation in another interventional study involving human participants or in the exclusion period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | At week 36
  Treatment failure is defined by any of the following in at least one eye:
  * new active, inflammatory chorioretinal or retinal vascular lesions;
  * worsening of Best Corrected Visual Acuity (BCVA) by>3 lines; Score from 20/10 (best vision) to 20/2400 (worst vision).
  * 2- step increase in anterior chamber cell grade and/or in vitreous haze relative to baseline. Anterior chamber cells scored from 0 (None) to 4+ (intense: fibrin or plastic aquerous) and Vitreous haze Scored from 0 (<1 cell in field) to +4 (>100 cells in field)
  * absence of steroid discontinuation between week 13 and week 19 (as per protocol)
  * or any additional immunosuppressive drug or injectable steroids

SECONDARY OUTCOMES:
Time to treatment failure | Up to week 55
Best corrected visual acuity | At week 4
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 8
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 12
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 16
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 20
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 24
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 30
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 36
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Best corrected visual acuity | At week 55
  Snellen score in each eye. Score from 20/10 (best vision) to 20/2400 (worst vision).
Anterior chamber cell grade in each eye | At week 4
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 8
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 12
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 16
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 20
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 24
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 30
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 36
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Anterior chamber cell grade in each eye | At week 55
  Score from 0 (None) to 4+ (intense: fibrin or plastic aqueous).
Vitreous haze grade in each eye. | At week 4
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 8
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 12
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 16
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 20
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 24
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 30
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 36
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Vitreous haze grade in each eye. | At week 55
  Nussenblatt score, Score from 0 (<1 cell in field) to +4 (>100 cells in field)
Central retinal thickness in each eye from baseline | At week 4
Central retinal thickness in each eye from baseline | At week 8
Central retinal thickness in each eye from baseline | At week 12
Central retinal thickness in each eye from baseline | At week 16
Central retinal thickness in each eye from baseline | At week 20
Central retinal thickness in each eye from baseline | At week 24
Central retinal thickness in each eye from baseline | At week 30
Central retinal thickness in each eye from baseline | At week 36
Central retinal thickness in each eye from baseline | At week 55
Proportion of patients with central macular thickness< 300 microns | At week 4
Proportion of patients with central macular thickness< 300 microns | At week 8
Proportion of patients with central macular thickness< 300 microns | At week 12
Proportion of patients with central macular thickness< 300 microns | At week 16
Proportion of patients with central macular thickness< 300 microns | At week 20
Proportion of patients with central macular thickness< 300 microns | At week 24
Proportion of patients with central macular thickness< 300 microns | At week 30
Proportion of patients with central macular thickness< 300 microns | At week 36
Proportion of patients with central macular thickness< 300 microns | At week 55
Time to optical coherence tomographic (OCT) evidence of macular edema in at least one eye | Up to week 55
National Eye Institute Visual Functioning Questionaire-25 (VFQ-25) composite score | At week 12
  Note after responses converted: 100=Best, 0=Worst possible score
National Eye Institute Visual Functioning Questionaire-25 (VFQ-25) composite score | At week 24
  Note after responses converted: 100=Best, 0=Worst possible score
National Eye Institute Visual Functioning Questionaire-25 (VFQ-25) composite score | At week 36
  Note after responses converted: 100=Best, 0=Worst possible score
Measures of corticosteroid sparing | Up to week 55
  Percent meeting targets [<0.1 mg/kg/day prednisone], mean change, mean dose at week 55, and cumulative dose
Cumulative incidence of relapse | Up to week 55
Number of relapses | Up to week 55
Number of clinical manifestations of underlying disease | Up to week 55
  Depending on the underlying disease
Frequency and severity of adverse events | Up to week 55
Treatment discontinuation | Up to week 55

IPD SHARING:
Plan to Share IPD: Undecided